CLINICAL TRIAL: NCT04370847
Title: Ultrasonography for Fluid Assessment in Parturients With Preeclampsia Undergoing Elective Cesarean Section Under Spinal Anesthesia
Brief Title: Ultrasonography for Fluid Assessment in Parturients With Preeclampsia Undergoing Cesarean Section
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.19.10.235
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Elective Cesarean Section; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Ultrasound (LUS) Examination: Ultrasonographic assessment of fluid status through scanning the lungs would be performed in all included patients
  Interventions: Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Procedure: Cesarean Delivery; Radiation: lung ultrasound scans; Other: Ultrasound Assessment of the Inferior Vena Cava; Other: Optic nerve sheath diameter; Drug: ringer acetate; Drug: Intravenous Ephedrine; Drug: Intravenous Syntocinon

INTERVENTIONS:
Procedure: Spinal Anesthesia — Performed at the L3-L4 or L4-L5 interspace using a 25-gauge spinal needle
Drug: Intrathecal Bupivacaine — Bupivacaine 12.5 mg (2.5 mL 0.5%) will be administered in the subarachnoid space
Drug: Intrathecal Fentanyl — Fentanyl 15 μg will be administered in the subarachnoid space
Procedure: Cesarean Delivery — Lower segment cesarean section using the Pfannenstiel incision
Radiation: lung ultrasound scans — lung ultrasound scans will be performed while the patient is in the supine position with left lateral tilt by 30 degrees using a 2-5 MHz curved array transducer. The echo comet score (ECS) which corresponds to the amount of EVLW will be obtained by the 28-rib interspaces technique. An increased amount of (EVLW) is diagnosed by multiple B-lines or 'comet tails' which are defined as discrete laser-like vertical hyperechoic reverberation artifacts that arise from the pleural line and extend to the bottom of the screen without fading and move synchronously with lung sliding. The sum of the B-lines found on each of the 28 chest-wall areas yields the ECS.
Other: Ultrasound Assessment of the Inferior Vena Cava — The IVC largest and smallest diameters will be measured proximal to the opening of the M-mode using s2-4 MHz transducer placed longitudinally in the subcostal region.
Other: Optic nerve sheath diameter — Optic nerve sheath diameter measurement will be conducted in two axes of transverse and oblique sagittal using a 12-4MHz linear array transducer. Depth of the optic nerve will be localized and marked at 3 mm behind the retinal and optic nerve junction transverse diameter of optic nerve sheath will be calculated. The reported ONSD corresponds to the mean of the four values obtained for each patient transverse and sagittal plane for both eyes.
Drug: ringer acetate — 1000 ml ringer acetate will be administered over 2 hours.
Drug: Intravenous Ephedrine — Intravenous ephedrine 3, 5, and 10 mg will be administered when Systolic blood pressure decreases below 120, 110, and 90 mmHg, respectively.
Drug: Intravenous Syntocinon — Immediately after delivery, syntocinon 10 IU will be added to the running crystalloid solution.

SUMMARY:
Preeclampsia is a multifocal syndrome reported in 2-8 % of pregnancies. It is diagnosed in the second half of pregnancy by two separate measurements of systolic blood pressure ≥140 mmHg and/or a diastolic blood pressure ≥ 90 mmHg in the same arm and proteinuria >300 mg in 24 h urine collection. The risk for serious complications such as pulmonary edema, cerebrovascular accidents, coagulopathy, and hemorrhage is 10 to 30 fold higher among parturients with severe preeclampsia.

Severe preeclampsia is defined by one or more of the following clinical features: severe hypertension (systolic arterial pressure 160 mmHg and/or diastolic arterial pressure 110 mmHg on more than one occasion at least 4 h apart while the patient is on bed rest, renal dysfunction (serum creatinine >1.1mg/dl or doubling of serum creatinine in the absence of another renal disease, platelet count less than <100,000 mm3, acute pulmonary edema, epigastric pain not responding to medical treatment, new-onset cerebral and visual manifestation, hemolysis, elevated liver enzymes and low platelet count syndrome (HELLP syndrome)

DETAILED DESCRIPTION:
Fluid resuscitation is a key determinant in the management of these parturients. Hypovolemia exacerbates organ failure, whereas volume overload results in pulmonary edema. In this setting, the use of noninvasive hemodynamic monitoring is associated with reduced mortality.

Point-of-care lung ultrasonography is used in many critical care settings as the initial diagnostic imaging study for patients with respiratory symptoms. It is highly sensitive for the diagnosis of pulmonary edema which may occur even without cardiomyopathy or heart failure.

The IVC is a highly compliant vessel that changes its diam¬eter in parallel with changes in blood volume and central venous pressure. Measurement of IVC diameter and col¬lapsibility index using ultrasound through a subcostal approach has been investigated in patients of various settings. The IVC-CI imaging technique may be used to assess the volume status in healthy parturients undergoing routine cesarean delivery as well as in high-risk parturients as preeclampsia.

Cerebral edema is predominantly vasogenic and may be related to the failure of cerebral autoregulation with subsequent hyperperfusion, blood-brain barrier disruption, and endothelial cell dysfunction. Ultrasonographic measurements of the optic nerve sheath diameter (ONSD) correlate with signs of raised ICP.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* 32 - 41 weeks gestational age.
* Preeclampsia: Blood Pressure ≥140/90 mmHg after 20 weeks' gestation and proteinuria ≥300 mg/24 hours or 1+ on urine dipstick
* Elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* Body mass index (BMI) ≥40 kg/m2.
* Significant cardiovascular disease
* Other obstetrical problems
* Other uteroplacental problems
* Abruption placenta.
* Already treated for acute lung pathology prior to enrollment.
* Contraindications to spinal anesthesia.
* INR >1.5 or PLT<100,000 /mm3.
* Women presenting in labor.
* Previous thoracic surgery.
* Previous ocular surgery
* Ocular trauma
* Glaucoma.
* Preoperative pulmonary disease:
* Increased serum creatinine level ≥1.1 mg/dL.

Ages: 19 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: The calculated sample size of the study will be 70 parturients at 5% level of significance and 80 % power, using the following formula:
  N= (Z1-α/2+Z1-β) ² σ1* σ2 / δ ² *2 Z1-α/2 = 1.96 Z1-β= 0.842 σ = SD (8, 9) δ = Expected difference to be detected before and after delivery (4). α = Level of acceptability of a false positive result (level of significance=0.05).
  β = Level of acceptability of a false negative result (0.20).
  1- β= power (0.80).The sample size will be increased to 100 parturients to compensate for protocol failures with incomplete data and to increase the power of the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic fluid assessment | Time frame:preoperative(baseline) and 2 hours after spinal anesthesia.
  Detection of change in overall number of B lines (ECS) by lung ultrasound

SECONDARY OUTCOMES:
Urine output | For 2 hours after spinal anesthesia
  total urine output at 2 hours after spinal anesthesia
Oliguria | For 2 hours after spinal anesthesia
  Incidence of oliguria defined as a total urine output <60 mL/hr
Ephedrine use | Intraoperative
  total ephedrine dose
Intraoperative bradycardia | Intraoperative
  Incidence of bradycardia (Heart rate <50 beats/minute)
Incidence of nausea and vomiting. | Intraoperative
  Incidence of nausea and/or vomiting as reported by the patient
Difference between overall number of b lines | baseline and 1hour post spinal
  difference between overall number of b lines preoperative(baseline) and at 1 hour after spinal anesthesia.
Inferior Vena Caval Diameters | Baseline, and at 1 and 2 hours post-spinal
  Maximum, minimum inferior vena cava diameters and inferior vena cava collapsibility index changes over time.
Difference between optic nerve sheath diameter | baseline,at 1hour and at 2 hours of spinal anesthesia.
  optic nerve sheath diameter changes over time.
Neonatal Apgar score | 5 min after delivery
  neonatal Apgar score to assess neonatal wellbeing at 5 min after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Aboelnour E Aboelnour, MD, Study Chair — Professor of Anesthesia and Surgical Intensive care,; Hanaa A Elbendary, MD, Study Director — Assistant Professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt.; Marwa L Abdo, MD, Study Director — Lecturer of Anesthesia and Surgical Intensive care,; Sherine A Bakrey, MD, Study Director — Lecturer of Anesthesia and Surgical Intensive care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available following publication for life-long.
Access Criteria: the data will be accessible to the investigators .and the PRS administrators with hiding the identifiers for the patients